CLINICAL TRIAL: NCT02538523
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia FX-635 on Low Back Pain
Brief Title: A Study to Evaluate the Effect of Low Level Laser Light on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_LBP_002
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Erchonia FX-635 (Active Comparator): The Erchonia FX-635 is made up of 3 independent 17 milliWatts (mW), 635 nanometer (nm) red laser diodes mounted in scanner devices with flexible arms positioned equidistant from each other.
  Interventions: Device: Erchonia FX-635
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia FX-635 but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia FX-635 — The Erchonia FX-635 is applied to the lower back and hips area for 20 minutes per treatment administration, 8 times across 4 weeks, 2 times per week.
  Arms: Erchonia FX-635
Device: Placebo Laser — The Placebo Laser is applied to the lower back and hips area for 20 minutes per treatment administration, 8 times across 4 weeks, 2 times per week.
  Arms: Placebo Laser

SUMMARY:
This study evaluates the effect of low level laser light therapy on reducing low back pain. Half of the participants will receive the actual treatment with the active laser and the other half of the participants will receive a placebo treatment with an inactive laser.

DETAILED DESCRIPTION:
Back pain is a common musculoskeletal disorder affecting 80% of people at some point in their lives. It is the second most common neurological ailment in the United States, second only to headache, and it is the most common cause of job-related disability and a leading contributor to missed work. Around $50 billion is spent in the U.S. each year to treat low back pain. Men and women are equally affected, with the most common age affected being between 30 and 50 years.

Most low back pain stems from benign musculoskeletal problems, referred to as non-specific low back pain, which is the etiology being evaluated in this study. It is caused by lumbar sprain or strain a stretch injury to the ligaments, tendons, and/or muscles of the low back.

Current mainstream treatment approaches for low back pain due to lumbar sprain strain focus on reducing pain and inflammation, including rest; oral and topical over-the-counter and prescription medications; local heat applications; massage and exercise. Alternative treatment options include acupuncture; chiropractic manipulation; biofeedback; traction; transcutaneous electrical nerve stimulation (TENS); and ultrasound. Surgical procedures are also a treatment option for low back pain, and although the outcomes are often poor and do not last, back surgery remains the 3rd most common form of surgery in the United States, with about 300,000 back surgeries performed annually.

Low Level Laser Therapy (LLLT) communicates information to the receptors on the membrane of the cell and mitochondrion (the enzymatic engine of the cell). This energetic information reaches the cell's DNA, which directly controls cell function. When the cells receive better information, they work better, as do the tissues they comprise, like bones, cartilage, tendons, ligaments, etc. In this way, LLLT promotes the healing and regeneration of damaged tissues, having both local effects on tissue function and also systemic effects carried throughout the body by the blood and acupuncture meridians. The key basic physiological effects of low level laser light include increased cell membrane polarization and permeability; Adenosine-5-triphosphate (ATP) production and respiratory chain activity; enzyme activity; collagen and epithelial production; capillary formation; macrophage (immune) activity; analgesic effects due to elevated endorphin production, electrolytic nerve blockage, and improved blood and lymph flow; anti-inflammatory effect due to improved circulation and accelerated tissue regeneration; and increased production of antioxidants. Of additional benefit is that light energy from low level lasers will only be absorbed by cells and tissues that are not functioning normally and has no effect on healthy cells.

Therefore, low level laser therapy has the potential benefit of providing an effective means of reducing low back pain that is simple, quick, non-invasive and side-effect free.

ELIGIBILITY:
Inclusion Criteria:

* Primary pain is in the lower back region bound between the lowest rib and the crease of the buttocks
* Low back pain is of musculoskeletal origin wherein the etiology is lumbar sprain or strain
* Diagnosis is based on positive supportive patient history, physical examination, medication use history and review of relevant records and diagnostic tests
* Low back pain is episodic chronic, defined as pain having occurred on at least 15 days of each of the preceding 3 months, with each individual episode having lasted at least 24 hours followed by a subsequent period of at least 24 hours without pain
* Self-reported Degree of Pain rating on the 0-100 Visual Analog Scale (VAS) scale of 40 or greater
* Subject is willing and able to refrain from consuming any over-the-counter or prescription medications, including herbal supplements for the relief of pain or inflammation, including muscle relaxants throughout study participation, except for the study pain relief medication
* Subject is willing and able to refrain from non-study procedure therapies for low back pain throughout study participation
* Primary language is English

Exclusion Criteria:

* Low back pain is undiagnosed, or has been diagnosed as in whole or in part due to mechanical, inflammatory: neoplastic, metabolic or psychosomatic origins
* Non-organic pain, defined as positive findings for 3 or more of the 5 signs in the 'Waddell's Signs of Inorganic Behavior' list
* Known herniated disc injury
* Known osteoporosis with compression fractures
* Osteoporosis defined as a Total SCORE on the Simple Calculated Osteoporosis Risk Estimation (SCORE) screening questionnaire of > 6, and a Dual-Energy X-ray Absorptiometry (DEXA) T-score ≤ -2.5
* Congenital deformity of the spine
* Current, active chronic pain disease
* Cancer or treatment for cancer in the past 6 months, including spinal cord tumors
* Use of the analgesics paracetamol, compound analgesics or topical analgesics within 7 days prior to treatment
* Use of the muscle relaxants cyclobenzaprine (Lexeril, Fexmid), diazepam (Valium) or meprobamate (Miltown®, Equinil®, Equagesic®, Meprospan®) within 30 days prior to treatment
* Use of the muscle relaxants Carisoprodol (Soma®, Sodol®, Soprodol®, Soridol®) or Metaxalone (Skelaxin, Robaxin) within 7 days prior to treatment
* Use of the antidepressants duloxetine (Cymbalta®, Effexor), amitriptyline, imipramine (Tofranil), clomipramine (Anafranil), nortriptyline (Pamelor), desipramine (Norpramin) or selective serotonin reuptake inhibitors (SSRIs) e.g. Paxil, paroxetine, fluoxetine (Prozac) initiated within 30 days prior to treatment
* Consumption of systemic corticosteroid therapy or narcotics within 30 days prior to treatment
* Local or epidural injection of corticosteroids in the back within 3 months prior to treatment
* Botulinum toxin (Botox®) injection for chronic low back pain within 4 months prior to treatment
* Active infection, wound or other external trauma to the treatment areas
* Prior surgery to the back or spine
* Medical, physical or other contraindications for, or sensitivity to, light therapy
* Pregnant, breast feeding, or planning pregnancy prior to study end
* Serious known mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years
* Mental illness/incompetence defined according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) definition and criteria
* Current and/or prior history of alcohol and/or other substance abuse, defined according to the DSM-V definition and criteria
* Developmental disability or cognitive impairment that may compromise study participation
* Involvement in litigation or receiving disability benefits related to the study parameters
* Participation in a clinical study or other type of research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Berry, DC, Principal Investigator
Locations (3):
- United States (3):
  - South Mountain Chiropractic Center, Chandler, Arizona
  - Quarneri Chiropractic Inc., San Mateo, California
  - Bloomfield Laser and Cosmetic Surgery Center, Bloomfield, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia FX-635 | Placebo Laser
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia FX-635 | Placebo Laser | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.41 (17.07) | 44.72 (13.02) | 45.47 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22 | 18 | 40
  Hispanic | 1 | 7 | 8
  African American | 3 | 2 | 5
  Asian | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
Duration of Low Back Pain [Mean (Standard Deviation); unit: months] — Population: One subject did not report duration of low back pain.
  months
    number analyzed (Participants) | 28 | 29 | 57
    (all) | 86.39 (80.46) | 92.74 (82.74) | 89.62 (80.87)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Whose Change in Pain Rating on the Visual Analog Scale (VAS) Met the Individual Subject Success Criteria
Description: The Visual Analog Scale (VAS) assesses level or degree of pain. It is a horizontal line anchored on the left by the label '0: no pain at all' and on the right by the label '100: worst pain imaginable'. The subject marks a location on the 0-100 line that appears to represent any level of pain he or she is experiencing at that time. This marking is measured with a 0 to 100 mm ruler and the number recorded. For the primary study outcome, the percent change in the VAS pain score recorded at baseline and endpoint is calculated for each subject. Individual subject success is a 30% or greater change in VAS pain scores. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A positive (+) percent change indicates an increase in pain level and is negative for individual subject success. Overall study success is defined as a 35% or greater difference between the proportion of individual successes in each treatment group.
Time Frame: Baseline and Two Months Post-Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Erchonia FX-635 | Placebo Laser
Number analyzed (Participants) | 29 | 29
Participants | 21 | 8
Statistical Analysis 1: Comparison: Erchonia FX-635 vs Placebo Laser; A Fischer's Exact Test for two independent proportions was conducted to compare the statistical significance of the 44.8% difference in proportion of successes between procedure groups at two-months post-procedure (study endpoint) relative to baseline evaluation; Test type: Superiority; p < 0.005, Fisher Exact

2. Secondary Outcome: Change in Total Score on the Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) is a 10-item questionnaire to quantify disability for acute or chronic low back pain. Each question is scored on a scale of 0 (least amount of disability) to 5 (most severe disability). The ODI is expressed as a percentage and calculated by dividing the summed score of all questions answered by the total possible score (that is dependent on how many questions are answered) and multiplying by 100. A total score of '0%' means no disability and a total score of '100%' means the maximum disability possible. Therefore, the higher the total score, the worse the disability, and the lesser the total score, the lesser the disability.
Time Frame: Baseline and Two Months Post-Procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erchonia FX-635 | Placebo Laser
Number analyzed (Participants) | 29 | 29
score on a scale | -12.27 (10.69) | -5.18 (12.64)
Statistical Analysis 1: Comparison: Erchonia FX-635 vs Placebo Laser; Differences is the statistical significance of change scores in ODI total score from study baseline to endpoint (two-months post-procedure) were evaluated by Analysis of Covariance (ANCOVA), with change from baseline to endpoint in ODI total score as the dependent variable, baseline ODI total score as the covariate and procedure group (Erchonia FX-635 or placebo laser) as a main effect; Test type: Superiority; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Erchonia FX-635 | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT02538523/Prot_SAP_000.pdf